CLINICAL TRIAL: NCT06949917
Title: Taste Perception,Oral Health Status and Selectied Salivary Hormones in Relation to Body Mass Index Among Agroup of Iraqi Adolescent Girls.
Brief Title: The Effect of Body Mass Index on Taste Perception,Salivary Hormones and Oral Health Status
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Basma abdulstar abdullah, Master student, Al-Mustansiriyah University
Other Study IDs: AL-Mustansiriyah University
Record Dates: First submitted 2025-04-14; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Oral Health; Tast Perference
MeSH Terms: interventions — Body Mass Index; Aging

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: body mass index for age — different body mass index according to age (normal weight,overweight,obeiece)

SUMMARY:
the goal of the study is to test the effect of body mass index on adolesent Iraqi student girls by measuring salivary hormones (ghrelin,leptin,resistin)and measuring oral health by plague index score() and taste perception score () 90 female subject will be enrolled in this study between 16-17 years old,30 subjects with normal body weight ,30 subject overweight ,and 30 subject with obeiece group catogerize by body mass index according to age.

the methed of the study is by taking Saliva sample from the subject , taste perception score and oral health measure.

ELIGIBILITY:
Inclusion Criteria:

* female
* 16-17 years old
* subject with no systemic diseas.

Exclusion Criteria:

* medically compressed patient
* patient with systemic disease

Ages: 16 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: female adolesent girls 16-17 years old
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
taste perception | taste perception for 90 subject of different body mass index
  taste perception scale score(1-6) to measure 90 subject
oral health status | oral health status will be measured for 90 subject of different body mass index.
  oral health status will be measured by plaque index score(1-3),gingival index score(1-3),and dental caries DMFT and DMFS .

SECONDARY OUTCOMES:
salivary ghrelin hormone | Baseline :salivary collection for ghrelin , salivary leptin and salivary resistin in AL least two hours fasting for different body mass index subject
  measure salivary ghrelin hormone of different body mass index of 90 subject to see if the body mass index effect on the salivary ghrelin hormon.
salivary leptin hormone | Baseline :salivary collection for ghrelin , salivary leptin and salivary resistin in AL least two hours fasting for different body mass index subject
  measure salivary leptin hormone of different body mass index of 90 subject to see if the body mass index effect on the salivary leptin hormon.
salivary resistin hormone | Baseline :salivary collection for ghrelin , salivary leptin and salivary resistin in AL least two hours fasting for different body mass index subject
  measure salivary resistin hormone of different body mass index of 90 subject to see if the body mass index effect on the salivary resistin hormon.